CLINICAL TRIAL: NCT06716684
Title: The Effect of Cognitive-Behavioral Approach Based Psychoeducation Program on Trait Anger and Anger Expression Styles of Nursing Students
Brief Title: Cognitive-Behavioral Approach and Anger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Berna Aktas, Assistant Professor, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Interventional trial
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Nursing Students; Psychoeducation; Anger
Keywords: Nursing Students; Psychoeducation; Cognitive Behavioral Approach; Anger; Anger Expression Style

STUDY DESIGN:
Intervention Model Description: Following recruitment, the nursing students were divided into a intervention and a control group by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the study, a 6-session psychoeducation programme on coping with anger was given to the intervention group.
  Interventions: Behavioral: Cognitive-Behavioral Approach Based Psychoeducation Program
- Control group (No Intervention): No intervention was applied to the control group in the study.

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Approach Based Psychoeducation Program — A 6 session cognitive-behavioral approach based psychoeducation program developed in line with the literature review is applied in the research. Group training sessions have been held once a week with each session 90 minutes on average. The techniques such as automatic thought recording, finding cognitive errors, thought-stopping, forming alternative thoughts, daydreaming, countdown, problem solving, role playing, modeling, deep breathing, relaxation exercises, summarizing, explaining, informing, homework were used in the sessions.
  Arms: Intervention group

SUMMARY:
A randomized controlled study was conducted to investigate the effects of a cognitive-behavioral approach-based psychoeducation program on nursing students' trait anger and anger expression styles.

DETAILED DESCRIPTION:
Anger, which is an emotion experienced by all people, is a natural and normal reaction that can occur depending on the interaction of the person with his/her environment. However, frequent anger can damage physical and mental health and can lead to violence and aggression. Anger is interpreted according to the way it is expressed and a person can express anger in different ways (anger-in, anger-out, anger-control). While anger-in and anger-out are negative behavioral reactions, anger control is an appropriate response. One of the groups that often experiences anger is nursing students. Students studying in the department of nursing are considered as the health workforce of tomorrow and both study in stressful environments and work in stressful environments. Anger is an emotion experienced as a reaction to stress among nursing students. The inability of students who do not have anger management skills to control their anger may negatively affect their approach to patients, relatives and teammates. Since negative expression of anger can have a negative impact on interpersonal relationships with others, it may hinder the development of working alliances between nursing students and patients. Students studying in the department of nursing graduate without adequate training on how to express their anger correctly. Anger coping programs for nursing students should primarily include the assessment of anger expression styles and provide techniques for expressing anger appropriately and coping with anger. This study aimed to investigate the effect of a psychoeducation program based on the cognitive-behavioral approach on nursing students' trait anger and anger expression style. The hypothesis that there was no difference between the intervention and control groups in terms of trait anger, anger-in, anger-out and anger control after the intervention were tested.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the study,
* Not to have participated in the training program on anger expression and management given by mental health professionals before,
* Not to have a psychiatric diagnosis-treatment history,
* Not to have hearing-vision problems,
* To be between the ages of 18-25,
* To have participated in at least four of the sessions,
* To get a high score from the Trait Anger Sub-scale compared to other students

Exclusion Criteria:

* Having previously attended a training program on anger expression and management given by mental health professionals
* Having a problem that prevents filling out the forms to be used in the research
* Having hearing or vision problems
* Being under 18 or over 25
* Having a history of psychiatric diagnosis and treatment
* Having not attended more than four sessions

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Trait anger and anger expression styles before intervention | Before the 6-week intervention was administered to students
  Students' trait anger and anger expression styles were assessed before the intervention. Trait Anger and Anger Expression Scale was used in the evaluation. Trait Anger and Anger Expression Scale: The 4-point Likert-type scale designed (1983) has a total of 34 questions. Turkish adaptation of this scale was made (1994). Ten questions in the scale question trait anger and twenty-four questions question anger expression styles. A score between 10-40 is obtained from the trait anger scale and between 8-32 from the other sub-scales (anger-in, anger-out and anger control). High scores from trait anger indicate that the level of anger is high, high scores from the anger control scale indicate that anger can be controlled, high scores on the anger-out subscale indicate that anger can be expressed externally, and high scores from the anger-in subscale indicate that anger is suppressed.

SECONDARY OUTCOMES:
Trait anger and anger expression styles after intervention | After the 6-week intervention was administered to students
  Students' trait anger and anger expression styles were assessed after the intervention. Trait Anger and Anger Expression Scale was used in the evaluation.

OTHER OUTCOMES:
Trait anger and anger expression styles three months after the intervention | Three months after the 6-week intervention was administered to students
  Trait anger and anger expression styles were assessed three months after the intervention. Trait Anger and Anger Expression Scale was used in the evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aktaş, PhD, Study Chair — Kafkas University Faculty of Health Sciences, Psychiatric Nursing Department
Locations (1):
- Kafkas University Faculty of Health Sciences, Department of Nursing, Psychiatric Nursing Department, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.